CLINICAL TRIAL: NCT02627443
Title: Phase 1 Dose Escalation and Expansion Cohort of Carboplatin and Gemcitabine With or Without M6620 (VX-970) in First or Second Recurrence Platinum-Sensitive Epithelial Ovarian, Peritoneal, and Fallopian Tube Cancer
Brief Title: Carboplatin, Gemcitabine Hydrochloride, and Berzosertib in Treating Patients With Recurrent and Metastatic Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-02064; NCI-2015-02064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1563; 9948 (Other: Dana-Farber - Harvard Cancer Center LAO); 9948 (Other: CTEP); N01CM00099 (NIH); P30CA015083 (NIH); UM1CA186686 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Fallopian Tube Carcinoma; Metastatic Ovarian Carcinoma; Metastatic Primary Peritoneal Carcinoma; Ovarian Endometrioid Tumor; Ovarian High Grade Serous Adenocarcinoma; Platinum-Sensitive Ovarian Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — berzosertib; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (carboplatin, gemcitabine hydrochloride, VX-970) (Experimental): Patients receive carboplatin IV over 30 minutes on day 1, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and berzosertib IV over 60 minutes on days 2 and 9. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Berzosertib; Drug: Carboplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of gemcitabine hydrochloride and berzosertib when given together with carboplatin in treating patients with ovarian, primary peritoneal, or fallopian tube cancer that has come back (recurrent) and has spread to other places in the body (metastatic). Chemotherapy drugs, such as carboplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Berzosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving berzosertib with chemotherapy (carboplatin and gemcitabine hydrochloride) may work better in treating patients with ovarian, primary peritoneal, or fallopian tube cancer compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess safety and tolerability of the combination therapy carboplatin, gemcitabine hydrochloride (gemcitabine), and berzosertib (M6620 [VX-970]) in adult women with platinum sensitive recurrent high grade serous or high grade endometrioid ovarian, primary peritoneal or fallopian tube cancer. (Phase I Dose Escalation/Safety Lead-in) II. Determine the dose of the triple therapy to be used in the dose expansion cohort of the study. (Phase I Dose Escalation/Safety Lead-in) III. Confirm the safety at the maximum tolerated dose (MTD) for the addition of M6620 (VX-970) to carboplatin and gemcitabine in first or second recurrence of platinum sensitive high grade serous or endometrioid ovarian, primary peritoneal or fallopian tube carcinoma. (Expansion Cohort)

SECONDARY OBJECTIVES:

I. To determine if the MTD for the combination of carboplatin, gemcitabine and M6620 (VX-970) improves the confirmed response rate in adult women with platinum sensitive recurrent high grade serous or high grade endometrioid ovarian, primary peritoneal or fallopian tube cancer.

II. To determine the impact of the MTD on overall survival (OS), duration of response, and progression-free survival (PFS).

INTEGRATED CORRELATIVE STUDY OBJECTIVES:

I. Collection of specimens for biomarker studies to provide preliminary proof of mechanism. Assess, in an exploratory fashion, whether the combination of gemcitabine and carboplatin activates the ATR/CHK1 pathway at achievable concentrations and also whether M6620 inhibits the activated pathway.

II. To determine whether increased deoxyribonucleic acid (DNA) damage as assessed by two different multiplex assays correlates with response to combination therapy with M6620 (VX-970).

III. To determine whether mutations in homologous recombination repair genes correlate with response to combination therapy with M6620 (VX-970).

IV. To ascertain modulation of ATR autophosphorylation and other pharmacodynamic readouts for ATR inhibition by M6620 (VX-970).

OUTLINE: This is a dose-escalation study of gemcitabine hydrochloride and berzosertib.

Patients receive carboplatin intravenously (IV) over 30 minutes on day 1, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and berzosertib IV over 60 minutes on days 2 and 9. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high grade serous or endometrioid ovarian, peritoneal or fallopian tube malignancy that is metastatic and for which curative measures do not exist. The histology can be confirmed from tissue that was taken at the time of diagnosis. A biopsy at the time of recurrence prior to enrollment on study is not required
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients enrolled in the expansion cohort will be required to have archival tumor tissue available for analysis and be willing to have a tumor biopsy at baseline (after registration and prior to starting study treatment), at cycle 1 day 2 and at cycle 2 day 2. Patients must have platinum sensitive disease and be in their first or second platinum sensitive recurrence. Platinum sensitive disease is defined as recurrence that occurred greater than six months after completion of their last line of platinum based therapy. No non-platinum regimens allowed; prior therapy with PARP inhibitors as well as bevacizumab is allowed
* No more than two prior platinum based regimens. One regimen is defined as the interval of treatment from start of platinum based doublet to finish of that treatment course for the initial therapy or for the recurrent disease episode. If the nonplatinum agent is altered due to any reason other than disease progression, it counts as one regimen. For example, if a patient started on carboplatin and paclitaxel but developed a taxol reaction and was switched to carboplatin and Abraxane, this counts as one prior regimen
* Children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Negative serum pregnancy test result for females of child bearing potential

  * Note: The effects of M6620 (VX-970) on the developing human fetus are unknown. For this reason and because deoxyribonucleic acid (DNA)-damage response (DDR) inhibitors as well as other therapeutic agents used in this trial may have teratogenic potential, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after completion of M6620 (VX-970) administration. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with platinum resistant disease or platinum sensitive disease that is past the first or second recurrence
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier, excluding alopecia. Patients with treatment related effects, such as peripheral neuropathy, that are grade 1 or less are eligible
* Prior exposure to gemcitabine
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX-970), carboplatin, gemcitabine or to these specific compounds
* M6620 (VX-970) is primarily metabolized by CYP3A4; therefore, concomitant administration with strong inhibitors or inducers of CYP3A4 should be avoided. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because M6620 (VX-970) as a DNA-damage response (DDR) inhibitor may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620 (VX-970), breastfeeding should be discontinued if the mother is treated with M6620 (VX-970). These potential risks also apply to the other agents used in this study, such as carboplatin and gemcitabine
* Patients with Li Fraumeni syndrome are excluded from the study as M6620 (VX-970) is a DDR inhibitor
* Addition of bevacizumab to the treatment in this study is not allowed; if the treating physician feels that the addition of bevacizumab is in the best interest of the patient, the patient should be treated with an FDA approved regimen outside of the present study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (phase I dose escalation) | Up to 28 days
  The MTD in this study will be defined as the highest safely tolerated dose, up to a maximum of dose level 4, where at most 1 out of six patients experience a dose limiting toxicity (DLT) with the next higher dose having at least 2 DLTs in 3 or more patients. Will be reported descriptively.
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Confirmed response rate | Up to 3 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
Overall survival (OS) | From study entry to death from any cause, assessed up to 3 years
  OS will be estimated using the Kaplan-Meier method.
Duration of response | From first documented date of confirmed response (complete response [CR] or partial response [PR]), to the date at which progression is first documented, up to 3 years
  The duration of confirmed responses will be assessed using the Kaplan-Meier method.
Progression free survival (PFS) | From registration to the first of either disease progression or death from any cause, up to 3 years
  Disease progression will be determined based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. PFS will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Changes in the frequency of marker inhibition | Baseline to up to 3 years
  Semi-quantitative data will be used to compare the data between the treatment arms using boxplots and descriptive statistics.
Correlation between deoxyribonucleic acid (DNA) damage markers and mutation data with clinical endpoints (i.e. response, PFS, OS) | Up to 3 years
  Statistical and graphical techniques will be used to explore these relationships. For time-to-event endpoints, we will use Cox proportional hazards models, and for response data we will use Logistic regression models. In addition, we will use Fisher's exact tests to test the association between categorical marker data and response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E Wahner Hendrickson, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (14):
- United States (14):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia